CLINICAL TRIAL: NCT06564077
Title: Effects of ELDOA in Patients With Upper Cross Syndrome
Brief Title: ELDOA's Effect in Upper Cross Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC 01937 Sundas Sultan
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Neck Pain
Keywords: Upper Cross Syndrome; ELDOA; pain
MeSH Terms: conditions — Neck Pain; Oculocerebral hypopigmentation syndrome type Preus; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eldoa technique with conventional therapy (Experimental): It is myofascial stretching technique of the cervical spine. Patients were asked to adopt desired position to target intervertebral segments. Breathing is also important factor in ELDOA stretch. Patients were instructed to not to hold or strain breathing through promoting diaphragmatic breathing.
  * Hot pack for 20 minutes
  * Strengthening exercises for deep neck flexors, rhomboids, serratus anterior, and lower trapezius (2 sets of 10 reps per day).
  * Stretching exercise for pectoralis muscle (20 sec hold,5 reps)
  Interventions: Other: Eldoa technique with conventional therapy
- conventional therapy (Active Comparator): * Hot pack for 20 minutes
  * Strengthening exercises for deep neck flexors, rhomboids, serratus anterior, and lower trapezius (2 sets of 10 reps per day).
  * Stretching exercise for pectoralis muscle (20 sec hold,5 reps)
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: Eldoa technique with conventional therapy — is myofascial stretching technique of the cervical spine. Patients were asked to adopt desired position to target intervertebral segments. Breathing is also important factor in ELDOA stretch. Patients were instructed to not to hold or strain breathing through promoting diaphragmatic breathing.
  * Hot pack for 20 minutes
  * Strengthening exercises for deep neck flexors, rhomboids, serratus anterior, and lower trapezius (2 sets of 10 reps per day).
  * Stretching exercise for pectoralis muscle (20 sec hold,5 reps)
  Arms: Eldoa technique with conventional therapy
Other: conventional therapy — * Hot pack for 20 minutes
  * Strengthening exercises for deep neck flexors, rhomboids, serratus anterior, and lower trapezius (2 sets of 10 reps per day).
  * Stretching exercise for pectoralis muscle (20 sec hold,5 reps)
  Arms: conventional therapy

SUMMARY:
The aim of this randomized clinical trial is to find the effects of ELDOA on decreasing pain ,kyphosis , improving range of motion and reducing disability

DETAILED DESCRIPTION:
Upper Cross Syndrome(UCS) is stress over the neck region due to poor posture and ergonomics, particularly sitting or standing. This syndrome can cause joint impairments, mainly targeting the atlanto-occipital joint, shoulder joint, C4-C5, and T4-T5 region . Poor posture can lead to stress on the cervico-thoracic or cervico-cranial junction. Upper crossed syndrome is given its name because an "X," in other words, a cross, can be drawn across the upper body. One arm of the cross indicates the muscles that are typically tight, and the other arm of the cross shows the muscles that are usually weak. Predominantly, the syndrome mainly occurs as a result of muscular imbalance that usually develops between tonic and weak muscles. This imbalance causes postural changes including forward head posture (FHP), hunching of the thoracic spine (rounded upper back), increased cervical lordosis, elevated and protracted shoulders, and scapular winging. The upper cross syndrome can lead to cervical and upper back pain and movement restrictions due to muscle imbalances, consequently causing poor quality of life.

ELDOA is a French acronym. The myofascial ELDOA technique was first described by Guy Voyer in 1979, which is also called LOADS (longitudinal osteoarticular de-coaptation stretching.It is based on active traction exercises for spacing the joint, fascial and spinal stretching by assuming a specific posture for 1 min. It targets spinal strengthening and decompression. ELDOA has originated from various treatment approaches and creates local and general effects. It allows decompression of zygopopheasal joints, more absorption of fluids in the disc, increase circulation, improve tone and end range. It also allows the correction of impaired posture, improving respiration and proprioceptive facilitation of the concerned segment. Myofascial tension induced between superior vertebra which is a wandering point and the inferior vertebrae which is a fixed point. Verbal cues are given to the subject for the encouragement goals and for maintaining proper position and not dropping a pose. Several conditions have been treated with ELDOA, including prolapsed intervertebral discs, piriformis syndrome, chronic low back pain, cervical radiculopathy, active trigger points, and forward head posture. Disc encryption existing at any level of the spine can be addressed through specific ELDOA poses.

The Rational of the present study is to determine the effects of ELDOA on decreasing pain, kyphosis, improving range of motion and reducing disability.

ELIGIBILITY:
Inclusion Criteria:

* Forward head posture (Measuring Tape used to record the tragus and wall distance in (cm) ,with considering the normative value 10 to 1055 cm in females and male respectively)
* Limited cervical range of motion (Flexion: less than 80◦, Extension: less than 70◦, Rotation: less than 90◦ both sides., Lateral flexion: less than 20◦)
* Kyphosis measure through flexi curve ruler
* Neck Pain more than 3 on NPRS scale

Exclusion Criteria:

* Participants having complaints of dizziness
* History of surgery or fracture
* Severe skin sensitization
* Cervical radiculopathy
* Trauma of upper extremity
* Malignancy of the upper limb or thorax
* Scoliosis

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NRPS) | two weeks
  The NPRS is a self-reported or clinician-administered measurement tool consisting of a numerical point scale with extreme anchors of "no pain" to "extreme pain". The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10 or 0-100 and can be administered in written or verbal form. The test-retest reliability for the NPRS has been demonstrated to be moderate to high, varying from 0.67 to 0.96. the NPRS has 0.79 to 0.95 convergent validity.
Neck disability index (NDI). | two weeks
  NDI is a patient completed, condition specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headache, concentration, work, driving, sleeping and recreation each section of 5 marks. Interpretation of this scale is as 0 score indicates no activity limitation and 5 score indicates complete activity limitation. Score ranges from 0 to 50 in which 0 indicates no disability and 50 means maximum disability. A higher score indicated a greater level of activity limitation
Inclinometer. | two weeks
  It is used to measure the cervical range of motion. Cervical spine in neutral position place one inclinometer on C7 spinous process and other over the top of head. adjust both inclinometer dial to 0. Patient perform ranges and record reading on both inclinometer. Mathematically difference between the 2 readings is range of motion.
Flexi curve ruler | two weeks
  A flexi curve ruler, is used for measuring a kyphotic index that is calculated as the width divided by the length of the thoracic curve, multiplied by 100. the evaluator mark the second and twelfth back vertebrae with a marker. All the measurements conduct in a relax standing position, that the subjects ask to put their weight between their legs and look directly to the front. After marking the intended points, the flexible ruler place on the spine in such a way that it takes shape of the selected area and there is no empty space between the ruler and the spine. Then, the marked points on the spine transfer to the ruler. At the end, the ruler carefully separate from the spine and place on the target paper, and the curves draw on the paper with a pencil and the target points specified. The distance between two points L and the depth of curvature H measure by the ruler and then measure through formula

CONTACTS AND LOCATIONS:
Overall Officials: maria Khalid, MSOMPT, Principal Investigator — Riphah International University
Locations (1):
- DHQ Hospital, Chak Six Hundred Twenty-four, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No